CLINICAL TRIAL: NCT04952831
Title: Utilization of Diffusion Magnetic Resonance Imaging (dMRI) in Evaluation of Spinal Cord Dysfunction and Prognosis in Patients With Cervical Spondylotic Myelopathy (CSM)
Brief Title: Diffusion MRI in Cervical Spondylotic Myelopathy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020408
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2020-09

CONDITIONS: Cervical Spondylotic Myelopathy
MeSH Terms: interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with mild CSM: mJOA score ≥15
  Interventions: Other: diffusion MRI (dMRI)
- Patients with moderate CSM: mJOA score 13~14
  Interventions: Other: diffusion MRI (dMRI)
- Patients with severe CSM: mJOA score ≤ 12
  Interventions: Other: diffusion MRI (dMRI)
- Controls: health volunteers
  Interventions: Other: diffusion MRI (dMRI)

INTERVENTIONS:
Other: diffusion MRI (dMRI) — All participants underwent dMRI scan at baseline

SUMMARY:
diffusion MRI in evaluates and predicts prognosis in CSM

DETAILED DESCRIPTION:
Cervical spondylotic myelopathy (CSM) is a spinal dysfunction disease common in the elderly population caused by cervical spine degeneration, spinal canal stenosis, and spinal cord compression. It may result in reduced quality of life or even disability. With the increased life expectancy of today's population, the incidence of CSM is increasing. Surgery is recommended to reduce compression of the spinal cord. However, due to individual differences and variations in spinal cord injury severity, the prognosis after surgery is often unpredictable. Therefore, proper evaluation of spinal cord function and prognosis prediction are important considerations for the clinical decision of whether to operate and selection of appropriate operation time. To achieve this goal, medical images are used to correctly evaluate the damage and recovery potential of neurons. Magnetic resonance imaging (MRI) provides spinal cord macrostructure details and can detect spinal cord damage. Clinically, conventional MRI is often used to confirm a CSM diagnosis and predict prognosis. However, MRI assessments, including increased signal intensity (ISI) and T1 hypo-intensity, might not be consistent with clinical manifestations or prognostic expectations.

Diffusion MRI (dMRI) enables early diagnoses and prognostic predictions due to its microstructure assessment advantages. The diffusion of water molecules is restricted due to structural barriers, such as axon membranes and myelin sheaths. Using the microscopic movement of water molecules, dMRI can detect microstructures indirectly using a model with specific underlying probability distribution function of diffusion. Three models are widely applied clinically: diffusion tensor imaging (DTI), diffusional kurtosis imaging (DKI), and neurite orientation dispersion and density imaging (NODDI). DTI assumes the diffusion distribution function to be Gaussian, DKI assumes it to be non-Gaussian, and NODDI assumes it to be multi-compartmental (intracellular pool, extracellular pool, and free water). Previous studies suggested the potential application value of DTI and DKI in patients with CSM; however, these models had limited specificity and were not sufficient to diagnose CSM in a clinical setting. Compared with DTI and DKI, NODDI has been shown to characterize spinal cord microstructure better.

ELIGIBILITY:
Inclusion Criteria:

* ages ranged 30-75
* compliance to MRI scan
* no MRI contraindication
* (Patients) clinical diagnosis of CSM and surgery in our hospital
* (Healthy controls) no spinal cord dysfunction

Exclusion Criteria:

* prior head or neck surgery or accompanying diseases with neurologic deficits and/or symptoms including multiple sclerosis, spinal cord injury, motor neuron disease, or spinal cord tumour
* images with motion artifact

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients come from the Peking University Third Hospital. Healthy volunteers come from online recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative neurologic improvement | 3-month, 6-month, 12-month, and 24-month
  Postoperative modified Japanese Orthopaedic Association (mJOA) and recovery rate (RR) at 3-month, 6-month, 12-month, and 24-month for patients
diagnosis of CSM | at baseline
  whether participants are diagnosed as CSM at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Huishu Yuan, Dr, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No